CLINICAL TRIAL: NCT01937923
Title: A Pre-Cellular Therapy Observational Study in Early Huntington's Disease
Acronym: PRE-CELL
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 455690; DR2A-05415 (Other Grant/Funding Number: CIRM)
Record Dates: First submitted 2013-08-26; First posted 2013-09-10 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Safety labs: Complete blood count, comprehensive metabolic panel, international normalized ration, partial thromboplastic time, thyroid stimulating hormone, urinalysis, HIV screen.
  Biomarkers: Brain-derived neurotrophic factor (BDNF) in cerebrospinal fluid (CSF) and Plasma, BDNF related and Huntington's Disease (HD) specific gene transcription markers in CSF and blood, Small molecule markers of HD in CSF and plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
This observational study will establish a clinical baseline and measure changes over time in movement, thinking, behavior, brain imaging, blood and spinal fluid markers in subjects with early stage Huntington's disease. Participants enrolled in this study may be eligible to participate in a future planned study of stem cell therapy for Huntington's Disease (HD).

In-person study visits occur at screening, baseline, and every 6 months thereafter for a minimum of 12 months, with interim phone call assessments.

DETAILED DESCRIPTION:
In PRE-CELL the investigators propose to enroll a cohort of early-stage HD patients in a prospective observational study designed to characterize clinical, neuro-imaging, laboratory and biomarker correlates of disease progression over 12-18 months. Subjects who complete a minimum of 12 months' participation in this trial will be candidates for enrollment in the future planned Phase 1 trial of intrastriatal delivery of mesenchymal stem cell (MSC)/Brain-derived neurotrophic factor (BDNF).

ELIGIBILITY:
Inclusion Criteria:

* Men or women age 18 and older, English speaking, able to give informed consent and comply with study procedures.
* HD diagnosis confirmed with genetic testing demonstrating CAG trinucleotide repeat length (CAGn) greater than 37
* Early stage HD with Total Functional Capacity (TFC) score of 9-13
* Demonstrable motor signs with a Unified Huntington's Disease Rating Scale (UHDRS) diagnostic confidence level of 4
* Must have a caregiver or informant able to give feedback about the participant and willing to report observations about subject on standardized forms.
* Subjects of child bearing potential must agree to adequate birth control measures including intrauterine device, hormone therapy, hormone rings or barrier methods including foams/gels AND condoms.

Exclusion Criteria:

* Very early disease without demonstrable motor signs (diagnostic confidence level < 4)
* Significant cognitive impairment or dementia as defined by Montreal Cognitive Assessment (MoCA) score < 12.
* Moderate or advanced disease with TFC < 9
* Concurrent active unstable psychiatric disease including history of suicide attempts within the last year, major personality or psychiatric disorders.
* History of concurrent serious medical illness such as HIV or current anti-retroviral treatment, cancer, major cardiac, pulmonary, immunological or other organ disease.
* History of coagulopathy, bleeding disorder, or concurrent use of blood thinners.
* History of brain tumor, serious traumatic brain injury with coma, or history of brain surgery.
* Any comorbid condition that presents an unacceptable health risk to the patient in the investigator's view
* Clinically significant laboratory test abnormalities, including full blood count, chemistry panel, liver function tests, Prothrombin time/international normalized ratio (PT/INR), lipid panel, electrocardiogram (EKG), or chest x-ray as judged by the investigator.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with safety or adherence to study requirements.
* History or documentation of contraindication for MRI brain scan, including the presence of pacemaker, neurostimulator, aneurysm clips, artificial heart valves, cochlear implants, metal fragments in the eyes, orbits or skin or any other known contraindication to MRI.
* Any significant MRI brain scan findings other than those characteristic of HD.
* Any contraindications to surgery or to the use of general anesthesia, including allergy.
* History of use of any investigational agent within 60 days prior to enrollment
* History of current or previous gene therapy or stem cell therapy.
* History of previous or current treatment with cytokines
* History of sensitivity to ganciclovir.
* Pregnant and/or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be primarily recruited from the Huntington's disease clinic in the University of California, Davis (UC Davis) department of neurology. We also plan to recruit participants from among northern California regional support groups, from letters to neurologists and psychiatrists who are treating patients with HD, from listing our study on clinical trials.gov, and at regional and national HD meeting presentations, and via print and video recordings on our website.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2013-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Rate of change from baseline in white matter volume on magnetic resonance imaging (MRI) brain scan. | Baseline and 12 or 18 months

SECONDARY OUTCOMES:
Rate of change from baseline on the UHDRS total motor score | Baseline and 12 or 18 months
Rate of change from baseline on the Total Functional Capacity score | Baseline and 12 or 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Vicki Wheelock, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Medical Center, Clinical Research Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tempkin T, DeCarli C, Scher L, Farias S, Duffy A., Fink K, Annett G, Brunberg J, Yarborough M, Hersch S, Stout J, Alyward E, Martin A, Kjer L, Swadell D, Nolta J, Wheelock V. PRE-CELL: A Pre-Cellular Observational Study in Early Huntington's Disease. Eight Annual Huntington's disease Clinical Research Symposium, Minneapolis MN, November 2014; Neurotherapeutics 2015;12(1): 263-284
- [Background] Wheelock V, Tempkin T, Duffy A, Martin A, Mooney L, Scher L, Farias S, Swadell D, DeCarli C, Brunberg J, Li C-S, Yarborough M, Dayananthan A, Stout J, Hersch S, Aylward E, Fink KD, Annett G and Nolta J. "PRE-CELL: Preparing for a future planned Phase 1 trial of genetically-modified stem cells over-expressing BDNF in patients with Huntington's disease." Ninth Annual Huntington's Disease Clinical Research Symposium (October 2015), Tampa FL
- [Background] Moscovitch-Lopatin M, DiFiglia M, Kegel-Gleason K, Ritch JJ, Rosenthal SJ, Sapp E, Wheelock V, Duffy A, Chopra V, Rosas HD, Hersch SM. "A Novel Translational Bioassay for Conformers of Mutant Huntingtin." Ninth Annual Huntington's Disease Clinical Research Symposium (October 2015), Tampa FL